CLINICAL TRIAL: NCT02412332
Title: Cell Therapy in Advanced Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Faculdade de Medicina do ABC (Other); IEP São Lucas - Instituto de Ensino e Pesquisa (Other); Hemocentro São Lucas (Unknown); CordCell (Unknown)
Responsible Party: Principal Investigator, João Tadeu Ribeiro Paes, Professor, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pacientes
Record Dates: First submitted 2015-03-24; First posted 2015-04-09 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: advanced COPD (stage III); Adult stem cells; Cell therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 - Control (No Intervention): The patients will be followed during the course of 12 months and evaluated regarding disease progression. No interventions will be performed other than conventional (in-course) treatment.
- Group 2 - BMMC (Experimental): Patients will be submitted to bone marrow harvesting. Bone marrow mononuclear cells (BMMC) will be obtained by Ficoll separation and returned to patients by systemic infusion (1x10^8 BMMC in 30 mL saline). Three patients will be submitted to Lung perfusion scintigraphy with technetium for cell engraftment evaluation.
  Interventions: Procedure: Bone marrow harvesting
- Group 3 - ASC (Experimental): Patients will be submitted to liposuction. The obtained fat tissue will be cultivated by 21 days and adipose-derived stem cell (ASC) will be returned to patients by systemic infusion (1x10^8 ASC in 30 mL saline). Three patients will be submitted to Lung perfusion scintigraphy with technetium for cell engraftment evaluation.
  Interventions: Procedure: Liposuction
- Group 4 - BMMC + ASC (Experimental): Patients will be submitted to liposuction and the obtained fat tissue will be cultivated by 21 days and adipose-derived stem cell (ASC) obtained. Patients will be submitted to bone marrow harvesting and bone marrow mononuclear cells (BMMC) will be obtained by Ficoll separation. BMMC and ASC will be returned to patients by systemic infusion (5x10^7 ASC + 5x10^7 BMMC in 30 mL saline). Three patients will be submitted to Lung perfusion scintigraphy with technetium for cell engraftment evaluation.
  Interventions: Procedure: Bone marrow harvesting; Procedure: Liposuction

INTERVENTIONS:
Procedure: Bone marrow harvesting — Approximately 200 mL of bone marrow will be surgically collect from the iliac crest (pelvis) of the patient under spinal anesthesia.
  Arms: Group 2 - BMMC; Group 4 - BMMC + ASC
Procedure: Liposuction — Approximately 50 mL of adipose tissue (fat) will be surgically collected from the abdominal region of the patient under spinal anesthesia.
  Arms: Group 3 - ASC; Group 4 - BMMC + ASC

SUMMARY:
The purpose of this study is to determine whether cell therapy with autologous adult stem cells (from bone marrow and/or fat) is safe in the treatment of advanced Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Pulmonary emphysema, within the spectrum of Chronic Obstructive Pulmonary Disease (COPD), can be described as the destruction of alveolar walls and enlargement of the airspaces distal to the terminal bronchioles, with inflammatory infiltrate and no detectable fibrosis. Despite significant advances resulting from the introduction of new therapeutic approaches, such as pulmonary rehabilitation, an effective and not only palliative clinical treatment is yet to be achieved. Surgical treatment, in turn, involves highly complex procedures and, in the case of lung transplantation, the shortage of donors. In this context, cell therapy with stem cells is presented as a promising therapeutic alternative with great potential for applicability. The main goal of this study is to evaluate the safety of the infusion of bone marrow mononuclear cells (BMMC), adipose-derived stem cells (ASC), separately or conjugated, in COPD patients. The sample will consist of 20 advanced COPD patients (grade 3 by GOLD criteria). Patients will be, by lot, divided into four distinct groups, namely: Group 1: Control; Group 2: Bone marrow mononuclear cells; Group 3 - Stem cells derived from adipose tissue and Group 4: bone marrow mononuclear cells and stem cells derived from adipose tissue. After the selection of patients, clinical and laboratory evaluation will be conducted (cardiology, laboratory examinations and tests to define the score of dyspnea). The cells used for the cell therapy will be obtained from the patient's own bone marrow or adipose tissue (autologous). The separation of the bone marrow mononuclear (BMMC) will be performed by centrifugation in density gradient (Ficoll), while stem cells derived from adipose tissue will be isolated by enzymatic digestion (collagenase) and cultivation. The infusion will be performed by a peripheral vein (brachial) after preparation, separation, expansion and quality control of the cells. The patients will be followed for a period of 12 months. It is expected that this clinical protocol will allow an expansion in knowledge about cell therapy in pulmonary diseases and represents a significant step towards the establishment of new therapeutic approaches in COPD treatment.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with persistent dyspnea in stage 2 or 3 of the dyspnea scale score;
* Eligibility for pulmonary rehabilitation program;
* No smoking or smoking cessation for at least 6 months.

Exclusion Criteria:

* Absence of emphysema on chest tomography;
* Pulmonary or extrapulmonary infection or active infection history in less than 3 months;
* History of coronary artery disease and/or severe ventricular dysfunction (ejection fraction <55%);
* Presence of pulmonary hypertension, ie, estimated systolic pulmonary artery pressure above 35 mmHg at transthoracic Doppler echocardiography;
* Patients in home oxygen therapy;
* Advanced renal failure (serum creatinine greater than 1.5 mg / dL) and liver failure CHILD B or C;
* Immunosuppressive or infectious diseases detected;
* Patients with known malignancies or collagen diseases;
* Psycho-social problems, drug and/or alcohol abuse and not obedient to the established medical protocol;
* No family acceptance;
* Pregnancy or at risk of pregnancy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Total Pulmonary Capacity | 12 months after procedure
  Assessed by whole body plethysmography, measured in liters.

SECONDARY OUTCOMES:
Pulmonary morphology | 9 months after procedure
  Chest x-ray
Pulmonary function | 12 months after procedure
  A composite measure of pulmonary capacity (volume), assessed by plethysmography and spirometry and composed of: Total Pulmonary Capacity (TPC), Forced Vital Capacity (FVC), Forced Expiratory Volume (FEV1) , FEV1/FVC, Forced Expiratory Fraction (FEF 25-75), Residual Volume (RV), TPC/RV and airway Resistance (R).

CONTACTS AND LOCATIONS:
Overall Officials: Selma D Squassoni, MD, Study Chair — Faculdade de Medicina do ABC; Ellie Fiss, MD, Study Chair — Faculdade de Medicina do ABC; Elíseo J Sekya, Study Chair — IEP São Lucas - Instituto de Ensino e Pesquisa; Adelson Alves, Dr, Study Chair — Hemocentro São Lucas; Andressa Forte, Study Chair — TechLife; Larissa C Zanutto, Study Chair — IEP São Lucas - Instituto de Ensino e Pesquisa
Locations (1):
- Laboratório de Genética e Terapia Celular - GenTe Cel, Assis, São Paulo, Brazil

REFERENCES:
- [Background] Stessuk T, Ruiz MA, Greco OT, Bilaqui A, Ribeiro-Paes MJ, Ribeiro-Paes JT. Phase I clinical trial of cell therapy in patients with advanced chronic obstructive pulmonary disease: follow-up of up to 3 years. Rev Bras Hematol Hemoter. 2013;35(5):352-7. doi: 10.5581/1516-8484.20130113. PMID 24255620
- [Background] Ribeiro-Paes JT, Bilaqui A, Greco OT, Ruiz MA, Marcelino MY, Stessuk T, de Faria CA, Lago MR. Unicentric study of cell therapy in chronic obstructive pulmonary disease/pulmonary emphysema. Int J Chron Obstruct Pulmon Dis. 2011 Jan 1;6:63-71. doi: 10.2147/COPD.S15292. PMID 21311694
- [Background] Ribeiro-Paes JT, Stessuk T, Marcelino M, Faria C, Marinelli T, Ribeiro-Paes MJ. A protocol proposition of cell therapy for the treatment of chronic obstructive pulmonary disease. Rev Port Pneumol. 2014 Mar-Apr;20(2):84-91. doi: 10.1016/j.rppneu.2013.06.008. Epub 2013 Nov 26. English, Portuguese. PMID 24287082